CLINICAL TRIAL: NCT01427621
Title: Effect of Combined Remote Ischemic Preconditioning and Postconditioning on Acute Pulmonary Injury in Patients Undergoing Valvular Heart Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 4-2009-0648
Record Dates: First submitted 2011-08-30; First posted 2011-09-01 (Estimated); Last update posted 2011-09-01 (Estimated); Status verified 2011-08

CONDITIONS: Heart Valve Diseases
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- RIPCcom group (Experimental)
  Interventions: Procedure: remote ischemic pre and postconditioning (RIPC)
- Control group (No Intervention)

INTERVENTIONS:
Procedure: remote ischemic pre and postconditioning (RIPC) — RIPCcom group: combined intervention of remote ischemic pre- and postconditioning consisted of three 10-minute cycles of right lower limb ischemia, which was induced with an automated cuff-inflator placed on the right upper leg and inflated to 250 mmHg, with an intervening 10 minute of reperfusion during which the cuff was deflated. This intervention were performed at 10 minutes after induction of anesthesia and then 10 min after weaning from CPB.
  Other Names: combined intervention of remote ischemic preconditioning and remote ischemic postconditioning.
  Arms: RIPCcom group

SUMMARY:
Pulmonary dysfunction after cardiac surgery with CPB remains to be a problem complicating the postoperative course of the patients. The investigators hypothesized that RIPCcom, combined intervention of remote ischemic preconditioning and remote ischemic postconditioning, would confer beneficial influence on inflammatory response and resultant postoperative pulmonary dysfunction after CPB in patients undergoing complex valvular heart surgery who are at increased risk of postoperative pulmonary dysfunction.The aim of this study was to evaluate the lung-protective effect of combined remote ischemic pre- and post-conditioning in patients undergoing complex valvular heart surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing valvular heart surgery.
* Age: 20~80.

Exclusion Criteria:

* Emergency operation.
* patients with peripheral vascular disease.
* Patients with a known history or clinical evidence of chronic obstructive pulmonary disease.
* Patients with hepatic or renal dysfunction
* Patients with acute myocardial infarction within 1 week before surgery

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2010-03; Primary Completion 2010-11 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Comparison of postoperative PaO2/FiO2 | at 10 minutes after anesthetic induction
  Comparison of postoperative PaO2/FiO2 between RIPCcom group and Control group.

CONTACTS AND LOCATIONS:
Overall Officials: Young-Lan Kwak, MD, Ph.D, Principal Investigator — Department of Anesthesiology and Pain Medicine, Severance Hospital, Yonsei University College of Medicine

REFERENCES:
- [Derived] Kim JC, Shim JK, Lee S, Yoo YC, Yang SY, Kwak YL. Effect of combined remote ischemic preconditioning and postconditioning on pulmonary function in valvular heart surgery. Chest. 2012 Aug;142(2):467-475. doi: 10.1378/chest.11-2246. PMID 22281799